CLINICAL TRIAL: NCT07351279
Title: " The Effect of Platelet Rich Fibrin On Sensitivity and Periodontal Pockets Distal to Second Molar After Surgical Extraction of Impacted Third Molar "
Brief Title: The Effect of Platelet Rich Fibrin On Sensitivity and Periodontal Pockets Distal to Second Molar After Surgical Extraction of Impacted Third Molar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Muhammad Umar Hayat, PGR OMFS( MDS), University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ERB167/2/02-07-2024/S1 ERB
Record Dates: First submitted 2026-01-11; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Third Molar Impaction; Surgical Extraction of Impacted Third Molars

STUDY DESIGN:
Intervention Model Description: Split mouth randomized, Controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case Group (Experimental): PRF placement in extraction socket
  Interventions: Other: Platelet rich fibrin
- Control Group (No Intervention): Surgical extraction without using PRF

INTERVENTIONS:
Other: Platelet rich fibrin — After surgical extraction of impacted mandibular 3rd molar PRF will be placed in extraction socket
  Other Names: PRF
  Arms: Case Group

SUMMARY:
Surgical extraction of impacted third molar is the most common surgical procedure performed in oral and maxillofacial surgery. The immediate post operative complications after 3rd molar surgery are pain, swelling and trismus while delayed post operative complications are mostly seen on the distal surface of second molar due to distal bone loss which include prolonged sensitivity due to increased periodontal pocket depth, gingival recession and root exposure.

When PRF clot is given in wound, it causes alterations of the cellular ratios in the wound blood clot, leading to replacement of blood cells with Platelets and growth factors stimulating all phases of healing which will improve the immidiate and delayed post operative complications The purpose of present study is to compare the clinical outcomes in the treatment of senstivity and periodontal pockets at the distal aspect of second molar following surgical extraction of impacted third molar using PRF or Blood clot alone.

DETAILED DESCRIPTION:
Impacted third molars distal to second molar are the cause of distal attachment loss leading to degradation of the interdental bone. This causes formation of periodontal pocket which leads to pericoronitis and further infection. If there is minimum or no distance between second and third molar, the loss of interdental bone leads to periodonto-pathogenic bacterial aggression. Partially impacted third molars are the active source of bacterial entry into the distal area of the second molar because of food retention and poor oral hygiene.

PRF is the second generation autologous platelet concentrate that is obtained from patient's own blood in simple and cost effective manner. PRF contains platelets, cytokines, leucocytes and circulating stem cells that are embedded in a heterogeneous fibrin matrix. These unique elements in PRF make it a good biomaterial that improves healing. The slow release of cytokines-vascular endothelial growth factor, transforming growth factor, Epidermal growth factor and platelet-derived growth factor-are the main components which play an important role in neo-angiogenesis and tissue repair which makes this particular material useful.

Platelet-Rich Fibrin (PRF), has potential to enhance soft and hard tissue healing However, the evidence surrounding its effectiveness in reduction of sensitivity and periodontal pockets remains inconclusive. Previous studies evaluating the use of PRF have reported contradictory results. While some have demonstrated a significant reduction in periodontal pocket depth and improved healing when PRF is applied to the extraction socket, others have found little to no difference when compared to surgical extraction without PRF placement. This inconsistency highlights the need for further investigation to clarify PRF's role in postoperative outcomes, particularly in relation to periodontal health distal to the second molar. In addition, many of the available studies on PRF in third molar extraction are limited by small sample sizes which reduces the statistical power and generalizability of their findings. Contradiction in their results are most probably due to small sample size Therefore study with larger sample size is required to validate previous results and offer more conclusive evidence Furthermore, there is a notable lack of research focusing on postoperative tooth sensitivity, which is a common patient complaint following third molar extraction. Existing literature has predominantly emphasized parameters such as pain, swelling, and periodontal pocket depth, while the effect of PRF on sensitivity remains largely unexplored. This represents a significant gap in research and patient-centered outcomes.

By assessing periodontal pocket depth, clinical attachment loss and sensitivity distal to the second molar with larger sample size, this study aims to offer a more integrated evaluation of PRF's effectiveness in third molar surgery

ELIGIBILITY:
Inclusion Criteria:

* Impacted third molar (as per Operational Definition) with fully erupted second molars bilaterally.
* Impacted Third molar with Class 2 and Level B according to Pell and Gregory's classification (Annexure B) with mesioangular or horizontal angulation of impaction
* Periodontal pocket depth > 4mm and Clinical attachment loss > 1mm at distal side of second molar
* Age 18-40 years, both genders.
* Patients who give informed consent.

Exclusion Criteria:

* Any Systemic Disease i.e. Uncontrolled Diabetes mellitus, Uncontrolled hypertension, Ischemic heart disease, bleeding disorders, Autoimmune diseases or immunocompromised patients
* Decayed or recommended for extraction second molars on either side.
* Allergic to Amoxicillin to standardize Antibiotic therapy protocol.
* Untreated periodontal condition.
* Inability to follow up.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Periodontal Pocket Depth | From Enrollment to end of treatment at 03 months
  Periodontal pocket depth will be measured as a distance between gingival margin and base of the periodontal pocket in millimeters by Williams periodontal probe .
Senstivity | from Enrollment to end of treatment at 03 months
  Response of patient elicited by painful stimulus i.e Tactile stimulus which is characteristically of short duration will be measured by Tactile method i.e. scratching the distal surface of second molar at cemento-enamel junction with dental explorer on Numeric scale with values from 0 to 10, 0 being the least/no sensitivity and 10 being the worst
Clinical attachment loss | From Enrollment to end of treatment at 03 months
  Clinical attachment loss will be measured as a distance between cemento-enamel junction of second molar to the base of periodontal pocket in millimeters by williams periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- Allama Iqbal Medical College/ Jinnah Hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Tadić, A., Bajkin, B., Mijatov, I., Mirnić, J., Vukoje, K., Sokač, M. And Vukelić, D., 2023. Influence of L-PRF topical application on bone tissue healing after surgical extraction of impacted mandibular third molars: A randomized split-mouth clinical study. Applied Sciences, 13, 4823.
- [Background] Sybil D, Sawai M, Faisal M, Singh S, Jain V. Platelet-Rich Fibrin for Hard- and Soft-Tissue Healing in Mandibular Third Molar Extraction Socket. Ann Maxillofac Surg. 2020 Jan-Jun;10(1):102-107. doi: 10.4103/ams.ams_228_19. Epub 2020 Jun 8. PMID 32855924
- [Background] Swetha Bhat, B., Periasamy, S. And Arun, M., 2021. Incidence of residual periodontal defects distal to second molar due to a mesioangular mandibular impacted third molar. International Journal of Dentistry and Oral Science, 8(7), pp. 3119-3123.
- [Background] Roy, I.D., Saxena, V., Babu, B.K.N. and Perumal, S.J., 2021. Efficacy of platelet-rich fibrin on pain, edema, and healing in mandibular third molar surgery: A split-mouth randomized study. Journal of Dental Defence Section, 15, pp. 21-30.
- [Background] Rocha MOC, Cruz AACF, Santos DO, Douglas-DE-Oliveira DW, Flecha OD, Goncalves PF. Sensitivity and specificity of assessment scales of dentin hypersensitivity - an accuracy study. Braz Oral Res. 2020 May 8;34:e043. doi: 10.1590/1807-3107bor-2020.vol34.0043. PMID 32401933
- [Background] Malhotra A, Kapur I, Das D, Sharma A, Gupta M, Kumar M. Comparative evaluation of bone regeneration with platelet-rich fibrin in mandibular third molar extraction socket: A randomized split-mouth study. Natl J Maxillofac Surg. 2020 Jul-Dec;11(2):241-247. doi: 10.4103/njms.NJMS_50_19. Epub 2020 Dec 16. PMID 33897188
- [Background] Lam, C.P., Nguyen, T.B.N. and Nguyen, T.B.L., 2023. Effect of platelet-rich fibrin on soft tissue, periodontal pocket healing, and alveolar bone height after third molar surgery: A randomized clinical trial. Scholars Journal of Dental Sciences, 10(7), pp. 121-127.
- [Background] Gasparro R, Sammartino G, Mariniello M, di Lauro AE, Spagnuolo G, Marenzi G. Treatment of periodontal pockets at the distal aspect of mandibular second molar after surgical removal of impacted third molar and application of L-PRF: a split-mouth randomized clinical trial. Quintessence Int. 2020;51(3):204-211. doi: 10.3290/j.qi.a43947. PMID 32020130
- [Background] Castro AB, Meschi N, Temmerman A, Pinto N, Lambrechts P, Teughels W, Quirynen M. Regenerative potential of leucocyte- and platelet-rich fibrin. Part A: intra-bony defects, furcation defects and periodontal plastic surgery. A systematic review and meta-analysis. J Clin Periodontol. 2017 Jan;44(1):67-82. doi: 10.1111/jcpe.12643. Epub 2016 Nov 24. PMID 27783851
- [Background] Bhujbal, R., Veerabhadrappa, S.K., Yadav, S., Chappi, M. And Patil, V., 2020. Evaluation of platelet-rich fibrin and platelet-rich plasma in impacted mandibular third molar extraction socket healing and bone regeneration: A split-mouth comparative study. European Journal of General Dentistry, 9, pp. 96-102.
- [Background] Abad CE, Sanz-Sanchez I, Serrano V, Sanz Esporrin J, Sanz-Martin I, Sanz M. Efficacy of the application of leukocyte and platelet-rich fibrin (L-PRF) on alveolar ridge preservation. A randomized controlled clinical trial. Clin Implant Dent Relat Res. 2023 Jun;25(3):592-604. doi: 10.1111/cid.13208. Epub 2023 Apr 23. PMID 37088697